CLINICAL TRIAL: NCT01917097
Title: Bradycardia Following Intraoperative Administration of Dexmedetomidine
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00524
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Tonsillectomy; Adenotonsillectomy
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dexmedetomidine patients: Patients that received dexmedetomidine during their surgery.
  Interventions: Drug: Dexmedetomidine
- No Dexmedetomidine: Patients that didn't receive dexmedetomidine during surgery.

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Groups: Dexmedetomidine patients

SUMMARY:
This is a retrospective chart review to evaluate the postoperative course of all pediatric patients admitted to the hospital following adenotonsillectomy over the past 24 months to evaluate the incidence of bradycardia in children who received dexmedetomidine intraoperatively and identify confounding factors which may be precipitating the bradycardia or potentiating the negative chronotropic effects of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing adenontonsillectomy or tonsillectomy during 2011 and 2012.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having ENT surgery at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Bradycardia | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States